CLINICAL TRIAL: NCT00852319
Title: Interpregnancy Care Project-Mississippi
Brief Title: Interpregnancy Care Project-Mississippi (IPC-M)
Acronym: IPC-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Mississippi State Department of Health (Other Government); Federally Qualified Community Health Centers (Unknown)
Responsible Party: Principal Investigator, Glen Graves, Professor, University of Mississippi Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-0017
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Premature Birth
Keywords: Interpregnancy Care; Preconceptual Care; Premature Birth; Preterm Delivery
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Central Mississippi group (Experimental): Participants from central Mississippi are provided with 24 months of interpregnancy care. The results from this arm are compared to a historical control group (who were not given interpregnancy care) from the same geographical area in Mississippi.
  Interventions: Behavioral: Interpregnancy Care
- Mississippi Delta group (Experimental): Participants from 18 counties of the Mississippi delta are provided with 24 months of interpregnancy care. The results from this arm are compared to a historical control group (who were not given interpregnancy care) from the same geographical area in Mississippi.
  Interventions: Behavioral: Interpregnancy Care

INTERVENTIONS:
Behavioral: Interpregnancy Care — The intervention package includes: 1) Creation of an individualized interpregnancy care plan based on assessments of risks for subsequent poor pregnancy outcomes; 2) Basic dental care and provision of primary health care services for 24 months; 3) Assistance in achieving a woman's desire for subsequent pregnancies and her need for optimum child spacing (ideally at least 18 months); 4) Provision of appropriate social services and community outreach in each woman's community.
  Arms: Central Mississippi group
Behavioral: Interpregnancy Care — The intervention package includes: 1) Creation of an individualized interpregnancy care plan based on assessments of risks for subsequent poor pregnancy outcomes; 2) Basic dental care and provision of primary health care services for 24 months; 3) Assistance in achieving a woman's desire for subsequent pregnancies and her need for optimum child spacing (ideally at least 18 months); 4) Provision of appropriate social services and community outreach in each woman's community.
  Arms: Mississippi Delta group

SUMMARY:
The IPC program will enroll women who deliver Very Low Birth Weight babies (stillborn or liveborn) at University of Mississippi Medical Center and women who have Very Low Birth Weight babies that receive treatment in the Neonatal Intensive Care Unit at University of Mississippi Medical Center and provide each woman with 24 months of funded comprehensive, integrated, primary health care services (including family planning, social services, general medical services,and basic dental care), and enhanced case management. The services will be community-based (via UMC Clinics, community health centers, and outreach programs) and will be provided by a multidisciplinary team of physicians, nurses, social workers, case managers, and Resource Mothers/Resource Workers. At the end of project follow-up, we will evaluate the success of the program in terms of improvement of general health status of enrolled women, and subsequent reproductive health outcomes (i.e., achieving reproductive intentions, intendedness and spacing of subsequent pregnancies, birth weight distribution of subsequent pregnancies) and cost of delivery services compared to reproductive health outcomes in the project's control population.

DETAILED DESCRIPTION:
In the United States, Low Birth Weight (LBW; less than 2500 grams) delivery is the leading cause of infant mortality for African Americans. In addition, Very Low Birth Weight (VLBW; less than 1500 grams) deliveries frequently result in severe chronic health problems and lifelong disability in the surviving children. The racial disparity in infant mortality between African Americans and Caucasians is widening throughout the United States. Since Mississippi is the only state in the country with almost 50 percent of births to African Americans, the impact on Mississippi is dramatic. Recent research has focused on fetal origins of adult chronic diseases such as diabetes and hypertension. These findings confirm that poor pregnancy outcomes such as VLBW infants are often trans-generational problems. They are more common among women in poor health who lack continuous access to primary health care.

The best clinical predictor of a woman's delivery of a VLBW infant is her history of a previous VLBW delivery. The base line rate of very low birth weight for the general population is 1.5 percent of live births. After the first VLBW delivery, African American women have a 13.4 percent chance of another VLBW delivery. These figures are doubled in the case of teen pregnancies and progressively rise with each additional VLBW delivery. Mississippi has approximately 40,000 births per year; less than 2.5 percent (800) of these pregnancies result in 50 percent of infant deaths.

In Mississippi, Medicaid coverage is available to many women during their pregnancies, including a subset of women who do not financially qualify for Medicaid outside of pregnancy. The majority of these women lose Medicaid eligibility approximately 60 days after delivery; therefore, they do not have access to primary care resources. It appears that the strategy that offers the greatest potential for increasing a high risk woman's chance of having a full term healthy baby is preconceptual and inter-conceptual care.

The proposed project identifies and enrolls women in the Interpregnancy Care Project (IPC) of Mississippi at discharge from the hospital following the delivery of a VLBW infant. The IPC program provides 24 months of primary, continuous health care, basic dental care, enhanced nurse case management, and community outreach via a resource mother or resource worker. Primary health care addresses key areas epidemiologically linked to a VLBW delivery including the following: 1) reproductive planning and short interpregnancy intervals; 2) poorly-controlled chronic diseases; 3) reproductive tract infections; 4) nutritional disorders and obesity; 5) depression and domestic violence; 6) substance abuse; and 7) periodontal disease and cavities. Peer group meetings are integrated with IPC health care visits. Resource mothers and resource workers focus on parenthood preparedness, safe housing, job skills training, and education in the form of home visits and telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* African American female
* Delivery of a VLBW (below 1500 grams) infant at University of Mississippi Medical Center; can be liveborn or stillborn
* Transfer of an otherwise-qualifying VLBW infant to University of Mississippi Medical Center within two months of birth
* Indigent or Medicaid-eligible during pregnancy
* Maternal residence in Hinds county or in one of the 18 delta counties in Mississippi's Federal Health Districts I, III, or V

Exclusion Criteria:

* Non-English speaking women
* Pregnant women are excluded because the program is designed to study the benefits of providing primary health care services during the interpregnancy period
* Women who are incarcerated or who are institutionally committed will be excluded because they will not be available to participate in the intervention package.

Ages: 13 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 264 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The average number of pregnancies conceived within 18 months of the index delivery. | The first 18 months the participant is enrolled in the study.

SECONDARY OUTCOMES:
The average number of adverse outcomes for pregnancies conceived within 18 months of the index delivery. Adverse outcomes include such events as preterm birth, miscarriage, stillbirth, low birth weight, and small size based upon gestational age. | The first 18 months the participants are enrolled in the program.
The health status of participants after participating in the study, highlighting the issues strongly associated with VLBW infants, such as diabetes, hypertension, and obesity. | Health status is assessed throughout the study.
The financial costs and feasibility of providing interpregnancy care to this high-risk population. | Over the course of this five-year study, the cost of providing interpregnancy care to this population will be compared to the general costs incurred by the control group that did not receive interpregnancy care.

CONTACTS AND LOCATIONS:
Overall Officials: Glen Graves, MD, Principal Investigator — University of Mississippi Medical Center
Locations (3):
- United States (3):
  - Mississippi State Department of Health, Jackson, Mississippi
  - Federally Qualified Community Health Centers, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi

REFERENCES:
- [Background] Dunlop AL, Dubin C, Raynor BD, Bugg GW Jr, Schmotzer B, Brann AW Jr. Interpregnancy primary care and social support for African-American women at risk for recurrent very-low-birthweight delivery: a pilot evaluation. Matern Child Health J. 2008 Jul;12(4):461-8. doi: 10.1007/s10995-007-0279-z. Epub 2007 Aug 22. PMID 17712612